CLINICAL TRIAL: NCT00960674
Title: Effects on Type 2 Diabetes by Tactile Massage Compared to Relaxation With Relaxation Tape
Brief Title: Tactile Massage in Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Per Wandell, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007/414-31/4
Record Dates: First submitted 2009-07-24; First posted 2009-08-18 (Estimated); Last update posted 2013-04-18 (Estimated); Status verified 2013-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tactile massage (Experimental): A gentle form of massage given once a week for three weeks
  Interventions: Procedure: Tactile massage
- Relaxation (Experimental): Relaxation (by the use of a CD with relaxation exercises used at least once a week for 10 weeks)
  Interventions: Behavioral: Relaxation

INTERVENTIONS:
Procedure: Tactile massage — Gentle massage given for one hour by specially educated massage therapists, usually registered nurses.
  Other Names: Relaxation
  Arms: Tactile massage
Behavioral: Relaxation — Relaxation by a CD with relaxation exercises, at least one hour per week for ten weeks
  Arms: Relaxation

SUMMARY:
Tactile massage is a gentle form of massage that probably exerts its effect through relaxation. In a pilot study of 11 subjects an effect on HbA1c of 0.8%-units was seen.

The study aimed at comparing the effect of tactile massage sessions for one hour given once a week for 10 weeks in comparison with relaxation through a relaxation CD performed once a week during 10 weeks. Primary outcome was HbA1c measured after completed intervention and after yet another 12 weeks. Secondary outcomes were quality of life by SF-36, other markers of metabolism (fasting glucose, insulin resistance by HOMA-model), inflammation (CRP, cytokines) and stress (cortisone, catecholamines).

DETAILED DESCRIPTION:
Effects of different relaxation techniques on metabolic control in type 2 diabetes have been described. A pilot study indicated an effect by tactile massage, a Swedish form of gentle massage given in sessions of around one hours and including treatment of the whole body in general, on metabolic control measured as HbA1c and on plasma corticosteroids.

The present study aimed at studying the effects in a randomized controlled study, with patients provided with a relaxation cd available at pharmacies in Sweden. Power calculations found that 20-25 subjects in each group would be sufficient to show effect on HbA1c (0.8% vs 0.3%), but that 45-50 subjects would be needed to show clinical relevant effect on quality of life.

Patients aged 35-75 years with type 2 diabetes and BMI 25-30 and HbA1c 6-8%-units (Swedish standard, corresponding to 7-9%-units in DCCT standard) from primary health care centres in Stockholm County were invited to participate, and was randomly assigned to tactile massage or relaxation groups.

Exclusion criteria was heart or renal failure, treatment with insulin, problems with Swedish language. Besides, only subjects of Swedish ethnicity were included in this first study, in order to refine results and avoid confusional results.

Examination with laboratory tests, body examination and questionnaire, including SF-36 and questions on smoking, dietary and physical activity habits, was performed before intervention, after the 10 weeks examination and after yet another 12 weeks. Urine sampling on catecholamines and corticosteroids was performed, and blood tests on HbA1c, fasting glucose, insulin, CRP, cytokines (TNF-alpha, IL-6), adiponectin, leptin, ghrelin.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* 35-75 years
* BMI 25-30, HbA1c (Swedish standard)
* Oral antidiabetic treatment

Exclusion Criteria:

* Heart failure
* Renal failure
* Insufficient knowledge in Swedish

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2007-08; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
HbA1c | 2008

SECONDARY OUTCOMES:
Quality of life by SF-36 | 2008

CONTACTS AND LOCATIONS:
Overall Officials: Per E Wändell, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Center for Family and Community Medicin, KI, Huddinge, Sweden